CLINICAL TRIAL: NCT05692648
Title: Effect of Repositioning Frequency on Bilirubin Level and Infant Comfort in Neonates Receiving Phototherapy
Brief Title: Effect of Repositioning Frequency Neonates Receiving Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sevinc Akkoyun, lecturer (Phd), Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/14489
Record Dates: First submitted 2022-12-31; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Bilirubinemia; Newborn Jaundice
Keywords: bilirubin; comfort; neonates; phototherapy; positioning
MeSH Terms: conditions — Hyperbilirubinemia; Jaundice, Neonatal | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: single-centered, single-blind, 3-arm, pretest-posttest parallel-group randomized controlled trial
Who Masked: Participant
Masking Description: single (participant, outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine position group (Experimental): These neonates were placed in supine position, fed every 2 hours in accordance with routine clinical practice, and then returned to supine position.
  Interventions: Behavioral: Supine position group
- Hourly position change group: (Experimental): Infants in this group were repositioned "every hour" based on the time of phototherapy initiation. Neonates were initially placed in supine position and then changed to the prone position. Infants were alternated between supine and prone positions every hour for 24 hours.
  Interventions: Behavioral: Hourly position change group
- Control Group (2-hour position change) (Other): Neonates in this group were repositioned every 2 hours as routine practice based on the time of phototherapy initiation.
  Interventions: Behavioral: Control Group (2-hour position change)

INTERVENTIONS:
Behavioral: Supine position group — These neonates were placed in supine position, fed every 2 hours in accordance with routine clinical practice, and then returned to supine position.
  Arms: Supine position group
Behavioral: Hourly position change group — Infants in this group were repositioned "every hour" based on the time of phototherapy initiation. Neonates were initially placed in supine position and then changed to the prone position. Infants were alternated between supine and prone positions every hour for 24 hours.
  Arms: Hourly position change group:
Behavioral: Control Group (2-hour position change) — Neonates in this group were repositioned every 2 hours as routine practice based on the time of phototherapy initiation. Phototherapy was started with neonates in supine position. In the second period, the neonate was placed in the prone position after routine feeding was performed.
  Arms: Control Group (2-hour position change)

SUMMARY:
Purpose: The present study was conducted to determine the effect of repositioning frequency during phototherapy on bilirubin level and neonates comfort.

Design and methods: This was a single-centered, single-blind, 3-arm, pretest-posttest parallel-group randomized controlled trial conducted in a neonatal intensive care unit. Participants were randomly assigned to one of three groups: Supine position group (n = 20), hourly position change group (n = 20), and control group (n = 20). The bilirubin level and comfort levels of the neonates were evaluated.

DETAILED DESCRIPTION:
Purpose: The present study was conducted to determine the effect of repositioning frequency during phototherapy on bilirubin level and neonates comfort.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 35-42 weeks
* birth weight of 2000 g or more
* indication for phototherapy
* no previous phototherapy,
* no medical diagnosis other than prenatal hyperbilirubinemia
* stable health status
* no clinical signs of dehydration
* transition to oral feeding, no sucking problems
* being at least 2 days old on the day of phototherapy

Exclusion Criteria:

* a sudden change in stability during phototherapy and
* phototherapy duration of less than 24 hours

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in bilirubin level | Baseline and 24 hours after phototherapy
  bilirubin level change
comfort level questionnaire | up to 24 hours
  comfort level change

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kücükoglu, professor, Study Director — Selcuk University; Fatma Tas Arslan, professor, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu/Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No